CLINICAL TRIAL: NCT06664307
Title: Evaluation of the Efficacy and Safety of Portal Pressure Gradient (PPG) Measurement Guided by Endoscopic Ultrasound (EUS) in the Therapeutic Algorithm of Patients with Liver Cirrhosis.
Acronym: GPP-USE
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Lourdes Grande Santamaría, ESPECIALISTA DE APARATO DIGESTIVO, Hospital Universitario Virgen Macarena
Other Study IDs: GPP-USE
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Portal Pressure Gradient (PPG) Measurement Guided by Endoscopic Ultrasound (EUS); Hepatic Cirrhosis
Keywords: Portal pressure gradient (PPG), endoscopic ultrasound (EUS) ,.the acute hemodynamic response
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients attending the hepatology clinic or hospitalized with a diagnosis of liver cirrhosis: All patients attending outpatient clinics or hospitalized with a diagnosis of viral etiology or alcohol-related liver cirrhosis will be evaluated for the indication of primary prophylaxis with NSBB according to Baveno VII guidelines.
  The choice of NSBB type was mainly based on clinical parameters, regardless of the presence of an acute hemodynamic response. In patients who did not show signs of circulatory dysfunction or refractory ascites, carvedilol was preferred, as it has been shown to be more potent in decreasing portal pressure. Carvedilol was initiated at a dose of 6.25 mg/day and, if tolerated, was subsequently increased to a target dose of 12.5 mg/day. Higher doses of carvedilol were only used in cases of concomitant hypertension. For propranolol users, the dose was progressively increased until the heart rate decreased to approximately 55 beats per minute. In patients with significant ascites, a maximum dose of 80 mg/day of propranolol was administered.

SUMMARY:
The development of Clinical significant PH (CSPH) is a major driver of complications. PPG is the strongest predictor of decompensation . The shortcomings of GPVH measurements and invasiveness has resulted in an area of unmet clinical need. Non-selective beta-blockers (NSBB) have demonstrated efficacy in reducing PH. However, this requires a second invasive procedure, and there is high interindividual variability in the hemodynamic response to NSBB. EUS-guided GPP measurement emerges as a more accurate, accessible and less invasive technique to potentially predict chronic hemodynamic response. The aim of this project is to assess the safety and efficacy of EUS-derived GPP measurement (EUS-GPP) in patients diagnosed with cirrhosis, to assess the acute hemodynamic response through EUS-derived GPP to intravenous propranolol administration in order to determine the patients who would benefit from NSBB treatment in primary prophylaxis to prevent decompensation using a strategy guided by EUS-GPP measurement.

DETAILED DESCRIPTION:
Liver cirrhosis is a progressive disease with a continuum of compensated to decompensated stages. The development of portal hypertension (PH) and fibrosis are the primary pathophysiological processes in this clinical course. Clinical significant PH (CSPH) is a major driver of complications such as ascites and variceal bleeding. PPG is the strongest predictor of decompensation with a negative predictive value of 90% for PPG < 10 mmHg. Non-selective beta-blockers (NSBB) have demonstrated efficacy in reducing PH and preventing variceal bleeding. The clinical efficacy of NSBB is based on a significant reduction in PPG, estimated by HVPG measurement. However, this requires a second invasive procedure, and there is high interindividual variability in the hemodynamic response to NSBB. Therefore, the development of tools to identify patients who are likely to benefit from beta-blockers is an unmet clinical need. In this regard, PPG measurement guided by EUS can potentially predict the chronic hemodynamic response, serving as a strategy to guide therapy and identify patients who can benefit from NSBB in a single hemodynamic study, substantially reducing the need for repeated measurements. The aim of this project is to assess the safety and efficacy of EUS-derived GPP measurement (EUS-GPP) in patients diagnosed with cirrhosis, to assess the acute hemodynamic response through EUS-derived GPP to intravenous propranolol administration in order to determine the patients who would benefit from NSBB treatment in primary prophylaxis to prevent decompensation using a strategy guided by EUS-GPP measurement.

The natural history of cirrhosis can be described as a continuum from a compensated phase to decompensation and liver failure, marked by the development of overt ascites (or pleural effusion with a serum ascites albumin gradient [>1.1 g/dl]), encephalopathy (West Haven grade >II), and variceal bleeding, with a rate of 5 to 7% per year. This decompensation results in higher mortality and a median survival of 2 years compared to 12 years in the compensated phase1.

The events defining decompensation are hepatic fibrosis and the development of portal hypertension as the main pathophysiological processes of this clinical course. It has been demonstrated that the hepatic venous pressure gradient (HVPG) is the strongest predictor of decompensation, with a negative predictive value of 90% for HVPG less than 10 mm Hg2.

Compensated cirrhosis can be divided into 2 stages, based on the absence or presence of clinically significant portal hypertension (CSPH). Clinically significant portal hypertension (CSPH) is the main driver of complications3-4 - such as the development of ascites or variceal bleeding. It is important to note that CSPH, diagnosed by a hepatic venous pressure gradient (HVPG) of ≥10 mmHg, may be present before the complications of portal hypertension develop.

In general, CSPH is present in around 50 to 60% of patients with compensated cirrhosis without varices5-6, while patients with varices typically have an HVPG of at least 10 mmHg3-4. Patients with an HVPG >12 mmHg are at risk of variceal bleeding7. The risk of hepatic decompensation and mortality increases at HVPG levels >16 mmHg8, and at >20 mmHg, there is a higher frequency of uncontrolled bleeding, early rebleeding, and bleeding-related death3-9-10.

Non-selective beta-blockers (NSBBs) have demonstrated their efficacy in reducing portal hypertension and their role in the primary and secondary prophylaxis of variceal bleeding in patients with cirrhosis. The reduction in hepatic venous pressure gradient by NSBBs is associated with a lower risk of variceal bleeding and ascites, along with other benefits including improvement in bacterial translocation and prevention of spontaneous bacterial peritonitis, which have positive effects on survival1,3,11,12,13,14,15.

Such treatment is highly effective, accessible, and can reduce the prevalence of HVPG and decompensation.

The clinical efficacy of NSBBs for preventing portal hypertension-related events largely relies on a significant decrease in the portal pressure gradient, i.e., the "response," estimated by measuring HVPG via hepatic vein catheterization. Reductions in HVPG of at least 10%-20% (depending on whether we consider primary or secondary prophylaxis) or below 12 mmHg indicate a chronic hemodynamic response to NSBB treatment associated with decreases in bleeding-related events, ascites, and portal hypertension, as well as improvements in survival16. However, assessing the HVPG response to NSBB treatment requires a second invasive procedure.

The main drawback of NSBBs is the significant interindividual variability in hemodynamic response, even within a specific stage of the disease; therefore, the development of tools to identify patients most likely to benefit from beta-blockade is an area of unmet clinical need. In this regard, measurements of HVPG before and after intravenous administration of an NSBB may help overcome these limitations and potentially predict chronic hemodynamic response. This approach could serve as a strategy to guide therapy and identify patients who may benefit from it in a single hemodynamic study, substantially reducing the need for repeated measurements17.

The prognostic role of an acute hemodynamic response to intravenous propranolol in primary18,19 and secondary prophylaxis19 has been evaluated by three previous studies, which have linked the value of acute response to predicting overall hepatic decompensation and subsequent decompensations in particular. These studies particularly highlight the relevance of assessing acute response as a tool for early risk stratification and estimating treatment efficacy during a single hemodynamic study, being more cost-effective and time-effective, as well as less invasive than two consecutive measurements of HVPG with and without NSBB treatment. Additionally, although the evolution of the underlying liver disease may also provide prognostic information and theoretically may strengthen the prognostic value of chronic hemodynamic response status20, it complicates the assessment of a potential benefit of NSBB therapy in the individual patient. This is particularly relevant in the context of treatment approaches guided by hemodynamic response, as applied in the PREDESCI study.

However, the shortcomings of HVPG measurements, such as invasiveness and cost, have raised the question of whether we can accurately identify CSPH through other modalities. Endoscopic ultrasound (EUS) enables comprehensive diagnosis and therapy in advanced liver disease. One of the techniques guided by EUS involves the measurement of the portal pressure gradient (PPG)21.

The determination of the hepatic venous pressure gradient (HVPG) allows for the assessment of portal hypertension and the issuance of an evolutionary risk based on its magnitude (Table 1). It is performed approximately and indirectly by interventional radiology, through catheterization and pressure measurement in the suprahepatic vein, and then inflating a balloon, assuming that the pressure obtained in this manner (wedged pressure) is present in the portal vein. The HVPG is the result of subtracting the suprahepatic vein pressure from the wedged pressure. HVPG is considered normal when it is less than 5 mm Hg. Subclinical portal hypertension exists if it is > 5 mm Hg and < 10 mm Hg, and clinically significant if it is >10 mm Hg. HVPG is the best parameter predicting prognosis in patients with chronic liver diseases22, establishing the risk of complications and mortality, the response to treatment with beta-blockers, to antiviral agents, as well as evaluating the risk of liver failure after surgery for hepatocellular carcinoma19,23. However, this technique is only available in a few centers, uses ionizing radiation, is invasive, and does not accurately determine the actual pressure in the portal vein, making it not useful in cases of presinusoidal portal hypertension19.

Endoscopic ultrasound allows for direct pressure measurements in the suprahepatic vein and the portal vein, providing an accurate measurement of the portal pressure gradient (PPG). Comparative studies in animal models have shown comparable values between simultaneous determination of HVPG by interventional radiology and ultrasound-guided endoscopy24. Preliminary studies in humans, particularly in cirrhotic patients, have demonstrated its safety and accuracy, enabling the measurement of PPG and liver biopsy to be performed in the same endoscopic session25,26,27,28,29. A prospective, observational, multicenter study is registered in Clinical Trials (NCT04668664), currently recruiting, evaluating the efficacy and safety of PPG measurement obtained by endoscopic ultrasound in cirrhotic patients referred for upper gastrointestinal endoscopy or endoscopic ultrasound. This approach allows for a simplified assessment of the benefits of NSBB during a single invasive procedure and advances personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced liver disease with an indication for primary prophylaxis with NSBBs

Exclusion Criteria:

- Age < 18 years. 2. Advanced stage hepatocellular carcinoma not eligible for curative treatment. 3. Pregnancy. 4. Esophageal stenosis. 5. INR > 1.5. 6. Platelets < 50,000 µL. 7. Ascites. 8. Patients with any contraindication for performing an upper gastrointestinal endoscopy.

9. Patients with contraindication to NSBB treatment. 10. Refusal to sign the informed consent form to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attending the hepatology clinic or hospitalized with a diagnosis of liver cirrhosis and an indication for primary prophylaxis with NSBBs will be prospectively and consecutively included
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
- Endoscopic ultrasound with determination of the portal venous pressure gradient using a 25G needle with adapted | 12 months
  The portal pressure gradient (PPG) is obtained via transgastric, ultrasound-guided intraparenchymal hepatic puncture using a 25G needle (EchoTip Insight, Cook Medical®) equipped with a pressure gauge. Measurements are obtained in mm Hg. A puncture is made in the middle hepatic vein, and three pressure determinations are taken, each lasting one minute. The lowest observed pressure is recorded, and the mean is calculated. Subsequently, the left branch of the portal vein is punctured, and three measurements are taken, each lasting one minute, and their mean is calculated. The PPG is obtained by subtracting the mean pressures in the portal vein from the mean pressures in the hepatic vein.
  The pressure gauge recording the pressures is always fixed in the same position for all pressure measurements, positioned at the level of the patient's venous axis.
  After the initial hemodynamic assessment, propranolol (0.15 mg/kg of body weight; aqueous solution of propranolol hydrochloride [1 mg/ml] st

CONTACTS AND LOCATIONS:
Overall Officials: RAFAELR R ROMERO CASTRO, DOCTOR, Study Director — SAS
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, SEVILLA, Spain

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make IPD available.

REFERENCES:
- [Derived] Romero-Castro R, Silva-Albarellos E, Grandes-Santamaria L, Carmona-Soria I, Jimenez-Garcia VA, Rodriguez-Tellez M, Caunedo-Alvarez A. Endoscopic ultrasound-guided portal pressure gradient assessment of acute hemodynamic response to intravenous propranolol. Endoscopy. 2026 Mar;58(S 01):E40-E41. doi: 10.1055/a-2764-4494. Epub 2026 Jan 13. No abstract available. PMID 41529708